CLINICAL TRIAL: NCT07019142
Title: Effects of High-fat Diet (HFD) on Small Intestinal Microbiome in Healthy Volunteers
Brief Title: High-fat Diet (HFD) and Small Intestinal Microbiome
Acronym: FATBOM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-02116
Record Dates: First submitted 2020-10-16; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Microbial Colonization; Small Intestinal Bacterial Overgrowth
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: 10 healthy volunteers with descriptive assessment of Primary endpoint
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HFD-challenge (Other): Luminal application of liquid fat
  Interventions: Dietary Supplement: HFD

INTERVENTIONS:
Dietary Supplement: HFD — Luminal challenge with standardized volume, amount, calories of fat

SUMMARY:
The investigators aim to characterize the upper small intestinal microbiome in healthy conditions in dependency on feeding condition (starved vs. high-fat-challenged) and diet (before and after 3 day high-fat-diet)

Primary outcome will be the maximum culturable bacteria (aerobic and anaerobic) in small intestinal luminal content during acute liquid-fat challenge before vs. after a short-term (3 day) high-fat-diet

In this pilot study, healthy volunteers will undergo i) an upper endoscopy for harvesting of small intestinal juice, mucosal biopsies and ii) blood withdrawal at baseline (starved) as well as during acute one-time high-fat luminal stimulation (within 3 hours after baseline) utilizing microbiological culture and 16S-RNA sequencing. The same procedure will be performed after 3 day high-fat-diet.

During endoscopy an acute luminal high-fat challenge which will be repeated after a short-term (3 day) high-fat diet

DETAILED DESCRIPTION:
Background: The small intestine represents the major site of lipid metabolism and absorption. Its microbiome has recently been demonstrated to regulate adaptive digestive and absorptive responses to dietary lipids in mice. The microbiome was thereby demonstrated to be a culprit to obesity development. In fact, high-fat diet (HFD) induced changes in the microbiome are most pronounced in the small intestine and transplantation of small bowel microbes from HFD conditions increased lipid absorption compared with low-fat-diet-derived microbes. In humans, HFD induced microbiota alterations has been demonstrated as dysbiosis in colonic and fecal flora9 but changes in the small intestinal microbiome before the onset of obesity have not been addressed so far. In HFD-associated obesity, an increased frequency of small intestinal bacterial overgrowth (SIBO)38 is observed in humans. SIBO so far has been defined as the presence of more than 105 CFU/ml of luminal aspirate or presence of colonic type bacteria determined by microbiological culture techniques5. Therefore, the current definition of SIBO has severe limitations. Specifically, this definition of SIBO is arbitrary, limited to luminal aspirate, aerobic bacteria and assessment in starved conditions. In clinical practice, SIBO is virtually never tested according to this definition. Therefore, it would be of great interest to investigate whether SIBO can be re-defined by investigating the dynamic behavior of the microbiota in the upper small intestine i) before (starved) and after HFD-stimulation and ii) by deep sequencing of 16S-RNA in luminal aspirate as well as biopsies (mucosa-associated compartment). The investigators will perform an observational case-control study in lean healthy volunteers applying an acute (one-time exposure) and short-term (3 day) HFD-challenge assessing duodenal juice and biopsies for quantity and quality of microbial consortia. This will help to define the acute response of the small intestinal microbiome to HFD and ultimately set the stage for a new definition of SIBO.

Moreover, HFD is known to modulate a) the bile-acid-pool and b) gut-derived hormones such as incretins as well as c) thyroid-hormone-status. Thus, impact of acute (one-time exposure) and short-term (3 day) high-fat-stimulation on serum concentration and composition of bile-acids, incretins and thyroid-stimulating-hormone (TSH) plus peripheral thyroid hormones will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Adults ≥18 years of age
* BMI between 18.5 and 25 kg/m2

Exclusion Criteria:

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product,
* Define drugs not allowed during the study or for specific periods of time prior to the administration of the test dose,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the study,
* Other clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* inability or unwillingness to provide blood samples and tissue samples (biopsies),
* Participants taking oral anticoagulant or with bleeding disorders who would be at much higher risk of bleeding after biopsy samples or who are contraindicated for an endoscopic examination,
* Uncertain diagnosis, non-resident patients and patients unable to give informed consent
* Patients that undergo chemotherapeutic treatment,
* Patients that have been under antibiotic therapy in the last 4 weeks,
* Pre-existing conditions that would distort results (e.g. SIBO, IBD, obesity, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Culturable bacteria | 3 days
  Maximum culturable bacteria (aerobic and anaerobic) in small intestinal luminal content during acute liquid-fat challenge before vs. after a short-term (3 day) high-fat-diet

CONTACTS AND LOCATIONS:
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
undecided